CLINICAL TRIAL: NCT05498922
Title: Effect of Mechanical Ventilation on Lung Development of Alveolar Stage
Status: Completed | Type: Observational
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-21-12
Record Dates: First submitted 2022-08-08; First posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-04

CONDITIONS: Mechanical Ventilation; Abnormal Lung Development
Keywords: Mechanical ventilation; Infant lung development

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Peak pressure when mechanical ventilation was switched around a reasonable range — The research protocol was approved by the Ethics Committee of Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, and written informed consents were obtained from all patients. After induction of anesthesia, Rb patients were transorally intubated and mechanically ventilated. The inspiratory time, ventilation rate, positive end-expiratory pressure, and oxygen concentration were set consistently among patients. When anesthesiologist switch the peak pressure around a reasonable range, indices including tidal volume, lung compliance, mean airway pressure on ventilator screen changed and were recorded when stable. All the ventilator setting parameters followed the guidance of mechanical ventilation in neonates and children (https://doi.org/10.1007/978-3-030-83738-9_8). All the anesthesia and ventilation performance were conducted by a fully qualified senior anesthesiologist to assure standardized and safe anesthesia, ventilation and operation procedure.

SUMMARY:
Human lung development begins at about 4-7 post-conception weeks (pcw), and lasts until 3 years after birth, which can be divided into five morphological stages. Alveolar stage is the last stage during which alveoli forms, contributing to the rapid increase of gas exchange surface. Alveolar stage spans from 36 pcw to age 3, so it could be influenced by external factors. Mechanical ventilation (MV) is not only an important rescue method for children with respiratory distress, but also an indispensable respiratory support for young children during surgeries. When ventilators expand alveoli by pushing gas into lung with positive pressure, it acts against physiological characteristics and was reported to cause ventilator-induced lung injury. However, for children under the age of 3 with healthy lung, whether and how MV affects lung development has not been clearly elucidated.

Pressure-controlled ventilation is the most common utilized ventilating method in neonates and infants, which adjusts peak inspiratory pressure (PIP) as needed to meet oxygenation and ventilation goal. Under same PIP, will tidal volume (Vt), mean airway pressure (MAP) be variable based largely on the patients' respiratory mechanics like lung compliance and airway resistance. Therefore, how previous MV affects the alveolar stage of lung development can be partly indicated by analyzing and comparing indices like Vt, MAP and lung compliance when collected under same ventilator settings in later MV.

Approved by the Ethics Committee of Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, and written informed consents obtained from all patients' guardians, this clinical research collected data from retinoblastoma patients under the age of 3, when undergoing transcatheter intracranial vascular embolization (TIVE), one of the main Rb treatments. These data can be divided into 3 categories,

* Patient characteristics, including age in days, gender, height and weight;
* Surgery information, including total number of operation and date of each operation;
* Mechanical ventilation information, including ventilation duration, Vt, lung compliance, MAP and PIP.

The respective contribution of PIP, operation number, age and body mass index (BMI) to Vt per BMI, pulmonary compliance and MAP were quantified as estimate with their significance (showed as p value), which were obtained by regression analysis.

More details are described in Detailed Description as follow.

DETAILED DESCRIPTION:
Human lung development begins in the early stage of intrauterine pregnancy, approximately 4-7 post-conception weeks (pcw), and lasts until 3 years after birth. It can be divided into five morphological stages, namely embryonic stage, pseudoglandular stage, canalicular stage, saccular stage and alveolar stage. Alveolar stage is the process of alveolar formation during which distal saccules subdivide into alveoli and fuse into capillary until completely surround it, contributing to the rapid increase of gas exchange surface. Alveolar stage spans from 36 pcw to 3 years of age, and thus could be influenced by external factors.

Mechanical ventilation (MV) is not only an important rescue method for critically ill children with respiratory distress, but also an indispensable respiratory support method for young children during pediatric surgeries. Different from spontaneous breathing which creates negative pressure in chest to bring in air, ventilators expand alveoli by pushing gas into lung with positive pressure. Therefore, no matter how ventilator nowadays has been optimized to provide breathing movement close to the natural breathing, it still acts against physiological characteristics and has been reported to cause ventilator-induced lung injury when giving respiratory support to both pediatric and adult patients in intensive care unit. However, for children under the age of 3 with healthy pulmonary system, whether and how MV affects the alveolar stage of lung development has not been clearly elucidated.

Pressure-controlled ventilation is the most common utilized ventilating method in neonates and infants, which adjusts peak inspiratory pressure (PIP) as needed to meet oxygenation and ventilation goal. Under same PIP, will tidal volume (Vt), mean airway pressure (MAP) be variable based largely on the patients' respiratory mechanics like lung compliance and airway resistance. Therefore, how previous MV affects the alveolar stage of lung development can be partly indicated by analyzing and comparing indices like Vt, MAP and lung compliance when collected under same ventilator settings in later MV.

Retinoblastoma (Rb) is a rare form of cancer that rapidly develops from the immature cells of a retina, the light-detecting tissue of the eye. It is the most common malignant cancer of the eye in children, and it is almost exclusively found in young children. Transcatheter intracranial vascular embolization (TIVE) is one of the main treatments for Rb, and to assure the smooth operation in pediatric children for their poor medical compliance, general anesthesia and MV are compulsory during TIVE. Given TIVE is usually performed time and time again to help attenuating cancer growth and delaying the diseased eye removal, we can infer the influence of MV on infant lung development by analyzing the contribution of MV operation number, which is also the TIVE operation times, to respiratory indices, with the premise that TIVE operation duration is nearly equal when it is operated by same clinical group.

Approved by the Ethics Committee of Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, and written informed consents obtained from all patients' guardians, this clinical research collected data from Rb patients under the age of 3, when undergoing TIVE. These data can be divided into 3 categories,

* Patient characteristics, including age in days, gender, height and weight;
* Surgery information, including total number of operation and date of each operation;
* Mechanical ventilation information, including ventilation duration, Vt, lung compliance, MAP and PIP under setting parameters recommended by the guidance of mechanical ventilation in neonates and children (https://doi.org/10.1007/978-3-030-83738-9_8).

The respective contribution of PIP, operation number, age and body mass index (BMI) to Vt per BMI, pulmonary compliance and MAP will be quantified as estimate with their significance (showed as p value), which can be obtained by regression analysis through statistical software SPSS Statistics. P < 0.05 is considered as statistically significant criteria.

ELIGIBILITY:
Inclusion Criteria:

* Age 0~3;
* History of full-term birth;
* Normal physical development in height and weight;
* Supine position during operation;

Exclusion Criteria:

* Congenital pulmonary dysplasia;
* Current or previous lung disease;
* Chest deformity;
* Additional interference to pulmonary breathing except MV during data collection;
* being involved in other clinical subjects.

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All recruited pediatric subjects were patients with retinoblastoma, of which girls constituted 47.61%. The youngest of patients was 4.5 months old and the oldest was 2.6 years old.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Tidal Volume (Vt) | an average of 5 minutes
  Vt is the quantity of gas delivered with each breath. In general, target tidal volumes in pediatrics range between 5 and 8 mL/kg of ideal body weight (IBW)
Pulmonary compliance | an average of 5 minutes
  pulmonary compliance is a measure of the lung's ability to stretch and expand. As an index of respiratory mechanics, it can indicate the stiffness of lung. For example, low pulmonary compliance is often seen in fibrosis.
Mean airway pressure (MAP) | an average of 5 minutes
  MAP typically refers to the mean pressure applied during positive-pressure mechanical ventilation. It correlates with alveolar ventilation, arterial oxygenation, hemodynamic performance, and barotrauma. It can also match the alveolar pressure if there is no difference between inspiratory and expiratory resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Lai Wang, Chief doctor, Principal Investigator — Department of Anesthesia, Shanghai Xinhua hospita
Locations (1):
- Department of Anesthesia, Shanghai Xinhua hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fernandes N., Chawla S. (2022) Mechanical Ventilation for Neonates. In: Sarnaik A.P., Venkataraman S.T., Kuch B.A. （eds） Mechanical Ventilation in Neonates and Children. Springer, Cham. https://doi.org/10.1007/978-3-030-83738-9_8
- See also: guidance of mechanical ventilation in neonates and children — http://doi.org/10.1007/978-3-030-83738-9_8

DOCUMENTS (2):
  • Study Protocol (2021-04-27): https://cdn.clinicaltrials.gov/large-docs/22/NCT05498922/Prot_000.pdf
  • Informed Consent Form (2021-04-27): https://cdn.clinicaltrials.gov/large-docs/22/NCT05498922/ICF_001.pdf